CLINICAL TRIAL: NCT01910363
Title: Comparison of Clinical Efficacy of Botulinum Neurotoxin Type A1 and A2 for Post-Stroke Lower Limb Spasticity: Phase 2/3
Brief Title: Study of a New Generation Botulinum Toxin A2NTX to Treat Spasticity After Stroke
Acronym: A2NTX
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Tokushima (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Principal Investigator, Ryuji Kaji, Professor and Chairman, Department of Neurology, University of Tokushima
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A1A2BONT; TU001 (Other Grant/Funding Number: Tokushima University)
Record Dates: First submitted 2013-07-18; First posted 2013-07-29 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Lower Limb Spasticity After Stroke
Keywords: poststroke spasticity; lower limb; botulinum toxin; A2
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A2NTX (Experimental): single intramuscular injection of 300 units of A2NTX, a purified low molecular weight (150 kDalton) botulinum toxin preparation of type A2
  Interventions: Drug: A2NTX
- BOTOX (Active Comparator): single intramuscular injection of 300 units of BOTOX®, a commercially available botulinum toxin preparation of type A1
  Interventions: Drug: BOTOX

INTERVENTIONS:
Drug: A2NTX — Intramuscular injection of the botulinum toxin preparation in 300 units (mouse LD50) into tibialis posterior and medial gastrocnemius muscles on the affected side.
  Other Names: A2NTX:low molecular weight (150kDalton) purified botulinum toxin type A2 preparation
  Arms: A2NTX
Drug: BOTOX — Intramuscular injection of the botulinum toxin preparation in 300 units (mouse LD50) into tibialis posterior and medial gastrocnemius muscles on the affected side.
  Other Names: BOTOX®:onabotulinumtoxinA (Allergan Co Ltd), commercially available botulinum toxin type A1
  Arms: BOTOX

SUMMARY:
To test the safety and efficacy of a new generation botulinum toxin preparation A2NTX for treating stroke patients with lower limb spasticity.

* we study the degree of spasticity in the ankle and knee joints, and walking speed in 30 patients with stroke before and after injecting 300 units of BOTOX or A2NTX in a blinded manner as for the patient, the physician, and the examiner.
* we also assess the safety of A2NTX and compare it to that of BOTOX.

ELIGIBILITY:
Inclusion Criteria:

* patients with lower limb spasticity after stroke
* duration more than 6 months
* Modified Ashworth Scale of ankle joint more than 2

Exclusion Criteria:

* patients with previous botulinum toxin injections to lower limbs
* patients with serious hepatic, renal or cardiac dysfunction
* patients with respiratory failure
* patients who cannot understand the instructions

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Ashworth Scale of the ankle joint | 30-60 days after injection
  Modified Ashworth Scale is measured at baseline, 30(27-33) days and 60 (56-63) days after injection. Area under curve of Modified Ashworth Scale changes at day 30 and day 60 after injection

SECONDARY OUTCOMES:
Change in Functional Independence Measure (FIM) | 30 days after injection

OTHER OUTCOMES:
Walking Speed for 3m | 30 days after injection
  Time required for a patient to stand up from sitting position in a chair of 50cm height and walk for 3m.
  If assistance is needed, the same method of assisting the patient is used throughout the study.
grasp power | 30 days after injection
  Grasping power of both upper limbs will be measure with a standard grasp measure device in kg units. Because injection is made into lower limbs, any decrease of grasp power will be assessed as the measure of unwanted spread of the toxin action.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokushima University Hospital, Tokushima, Tokushima, Japan

REFERENCES:
- [Derived] Kaji R. Clinical differences between A1 and A2 botulinum toxin subtypes. Toxicon. 2015 Dec 1;107(Pt A):85-8. doi: 10.1016/j.toxicon.2015.09.025. Epub 2015 Sep 21. PMID 26394198